CLINICAL TRIAL: NCT02050022
Title: Clinical Implementation and Outcomes Evaluation of Blood-Based Biomarkers for Chronic Obstructive Pulmonary Disease Management
Brief Title: Chronic Obstructive Pulmonary Disease Biomarker Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Centres of Excellence for Commercialization and Research (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Genome Quebec (Other); Providence Health & Services (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Don Sin, Dr. Don Sin, University of British Columbia
Other Study IDs: H11-00786
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Biomarkers; Genomics; Proteomics; Diagnostics; Prognostics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exacerbation: Patients experiencing acute exacerbation of COPD.
- Non-Exacerbation: COPD patients not experiencing acute exacerbation of COPD.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive disease that is characterized by loss of lung function, leading to breathlessness, poor quality of life, loss in productivity, and increased mortality. The World Health Organization estimates that COPD will be the third leading cause of death worldwide by 2020, accounting for more than 7 million deaths annually. COPD patients frequently experience 'lung attacks', during which breathlessness, coughing, and sputum production dramatically increase, leading to urgent office visits, emergency admissions and hospitalizations. Lung attacks reduce patient quality of life and cost the Canadian health care system nearly $4 billion dollars each year in direct and indirect costs. Lung attacks can be effectively managed if they are identified and treated early, but symptoms of a lung attack often overlap with those of other common conditions such as heart failure, pneumonia and even influenza. Because there are no tests that can separate lung attacks from these conditions, doctors struggle to accurately diagnose lung attacks at an early stage when drugs are most effective. This can lead to a delayed or even incorrect diagnosis and inappropriate treatment. This research will address this critical need. Our goal is to improve COPD patient care by developing new blood tests that will help identify patients who are in the early stages of a lung attack. Doctors will be able to use these tests to treat lung attacks at earlier stages than is currently possible. These blood tests will enable doctors to personalize management of COPD to meet the needs of the individual patient.

Hypothesis: New biomarker blood tests can be used to better identify and manage patients with COPD.

DETAILED DESCRIPTION:
An acute exacerbation of COPD (AECOPD) is defined as an acute event characterized by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication (in most cases to antibiotics and/or oral corticosteroids). In most cases of AECOPD, patients experience a gradual crescendo-like increase in shortness of breath, cough and purulent sputum production over days to weeks. At their peak, patients may experience extreme shortness of breath (sometimes described as "breathless paralysis") and uncontrollable paroxysms of cough and purulent sputum production. AECOPDs are complex physiological events. In 70-80% of cases, AECOPDs are precipitated by bacterial or viral respiratory tract infections. However, most patients who develop acute symptoms (e.g., runny nose, cough or fever) do not progress to AECOPDs and experience spontaneous resolution of their symptoms. Furthermore, many patients with COPD who do harbour pathogenic organisms in their airways do not develop AECOPD symptoms. Thus, other factors, including the host inflammatory response, likely play a role in the pathogenesis of AECOPDs. Prompt recognition and treatment of AECOPD during this prodromal period can abrogate full blown attacks. Thus by identifying and treating AECOPDs early on (in physicians' offices), emergency visits, hospitalizations, and even deaths can be significantly reduced. However, this is not easy as symptoms of AECOPD (especially early in their course) are non-specific and can easily be confused with other ailments such as heart failure, allergies, or even upper respiratory tract infections. Since there are no biochemical tests that clinicians can order to objectively confirm AECOPD, AECOPD can be missed entirely or misdiagnosed, leading to delayed treatments or in some cases to the wrong treatment, which may result in devastating consequences including respiratory failure, hospitalizations or even death. Once patients are in the full blown attack stage of AECOPD, treatments are only modestly helpful in relieving symptoms and hospitalization is often required to resolve them. The median duration of hospitalization for AECOPD in Canada is 10 days, followed by an average of 3 months of convalescence. Unfortunately, in most cases, full recovery is never achieved and patients continue to experience rapid decline in lung and physical function (compared to patients not hospitalized for AECOPD). The 3 year mortality rate following hospitalization is 50%, and hospitalizations and emergency visits are avoidable with earlier detection, diagnosis and treatment of AECOPD. Indeed, COPD is the leading cause of preventable hospitalization in Canada. However, without a simple blood test that primary care physicians (PCPs) can order in their offices, earlier diagnosis will not be feasible.

The primary objective of this study is to identify blood biomarkers that can diagnose AECOPD.

Following informed consent, blood samples will be collected from patients who are admitted for an exacerbation at day 1, 3 and 7 of their hospitalization and then at 30 days and 90 days post-hospitalization. Sputum samples will also be collected on the day of admission for AECOPD etiologic phenotyping. All patients receive standard anti-exacerbation care in hospital, including systemic corticosteroids and antibiotics and are followed both in and out of hospital by a transition team consisting of a nurse, physiotherapist and respiratory therapist with special expertise in COPD care.

Following informed consent of non-exacerbating patients, a blood sample will be collected which will be used as a comparison to the exacerbating patient samples.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* diagnosis of COPD
* patients admitted to the hospital for a COPD exacerbation OR attending the COPD clinic and not experiencing a COPD exacerbation

Exclusion Criteria:

* under 19 years of age
* patients seen in the COPD clinic who are experiencing an exacerbation

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exacerbation cohort: COPD patients who present in emergency or are admitted to Vancouver General Hospital or St. Paul's Hospital in Vancouver for a COPD exacerbation are approached for participation in the study.
  Non-exacerbation cohort: COPD patients who are seen in the hospital COPD clinic and are not experiencing an exacerbation are approached for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Exacerbation | Within 1 year
  Hospitalized and non-hospitalized exacerbations occurring within 1 year of hospital discharge from index hospitalization will be recorded. Non-hospitalized exacerbations will be defined by treatment with prednisone plus/minus antibiotics. Hospitalized exacerbations will be defined as a diagnosis of acute exacerbation of COPD at admission or at presentation to emergency.

CONTACTS AND LOCATIONS:
Overall Officials: Donald D Sin, MD, MPH, Principal Investigator — University of British Columbia, St. Paul's Hospital, James Hogg Research Centre
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Reid C, Haldar P, McCormick M, Haldar K, Kebadze T, Duvoix A, Lindblad K, Patel H, Rugman P, Dodson P, Jenkins M, Saunders M, Newbold P, Green RH, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Acute exacerbations of chronic obstructive pulmonary disease: identification of biologic clusters and their biomarkers. Am J Respir Crit Care Med. 2011 Sep 15;184(6):662-71. doi: 10.1164/rccm.201104-0597OC. PMID 21680942
- [Background] Aaron SD, Donaldson GC, Whitmore GA, Hurst JR, Ramsay T, Wedzicha JA. Time course and pattern of COPD exacerbation onset. Thorax. 2012 Mar;67(3):238-43. doi: 10.1136/thoraxjnl-2011-200768. Epub 2011 Oct 18. PMID 22008189
- [Background] Wilkinson TM, Donaldson GC, Hurst JR, Seemungal TA, Wedzicha JA. Early therapy improves outcomes of exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1298-303. doi: 10.1164/rccm.200310-1443OC. Epub 2004 Feb 27. PMID 14990395
- [Background] Sin DD, Man SF. Inhaled corticosteroids and survival in chronic obstructive pulmonary disease: does the dose matter? Eur Respir J. 2003 Feb;21(2):260-6. doi: 10.1183/09031936.03.00040803. PMID 12608439
- [Background] Sanchez M, Vellanky S, Herring J, Liang J, Jia H. Variations in Canadian rates of hospitalization for ambulatory care sensitive conditions. Healthc Q. 2008;11(4):20-2. doi: 10.12927/hcq.2008.20087. No abstract available. PMID 19066477
- [Background] Chapman KR, Bourbeau J, Rance L. The burden of COPD in Canada: results from the Confronting COPD survey. Respir Med. 2003 Mar;97 Suppl C:S23-31. doi: 10.1016/s0954-6111(03)80022-7. PMID 12647940
- [Background] Mittmann N, Kuramoto L, Seung SJ, Haddon JM, Bradley-Kennedy C, Fitzgerald JM. The cost of moderate and severe COPD exacerbations to the Canadian healthcare system. Respir Med. 2008 Mar;102(3):413-21. doi: 10.1016/j.rmed.2007.10.010. Epub 2007 Dec 20. PMID 18086519
- [Background] Sin DD, McAlister FA, Man SF, Anthonisen NR. Contemporary management of chronic obstructive pulmonary disease: scientific review. JAMA. 2003 Nov 5;290(17):2301-12. doi: 10.1001/jama.290.17.2301. PMID 14600189
- [Background] Malhotra S, Man SF, Sin DD. Emerging drugs for the treatment of chronic obstructive pulmonary disease. Expert Opin Emerg Drugs. 2006 May;11(2):275-91. doi: 10.1517/14728214.11.2.275. PMID 16634702
- [Background] Vestbo J, Anderson W, Coxson HO, Crim C, Dawber F, Edwards L, Hagan G, Knobil K, Lomas DA, MacNee W, Silverman EK, Tal-Singer R; ECLIPSE investigators. Evaluation of COPD Longitudinally to Identify Predictive Surrogate End-points (ECLIPSE). Eur Respir J. 2008 Apr;31(4):869-73. doi: 10.1183/09031936.00111707. Epub 2008 Jan 23. PMID 18216052
- [Background] Freue GV, Sasaki M, Meredith A, Gunther OP, Bergman A, Takhar M, Mui A, Balshaw RF, Ng RT, Opushneva N, Hollander Z, Li G, Borchers CH, Wilson-McManus J, McManus BM, Keown PA, McMaster WR; Genome Canada Biomarkers in Transplantation Group. Proteomic signatures in plasma during early acute renal allograft rejection. Mol Cell Proteomics. 2010 Sep;9(9):1954-67. doi: 10.1074/mcp.M110.000554. Epub 2010 May 25. PMID 20501940
- [Background] Gunther OP, Balshaw RF, Scherer A, Hollander Z, Mui A, Triche TJ, Freue GC, Li G, Ng RT, Wilson-McManus J, McMaster WR, McManus BM, Keown PA; Biomarkers in Transplantation Team. Functional genomic analysis of peripheral blood during early acute renal allograft rejection. Transplantation. 2009 Oct 15;88(7):942-51. doi: 10.1097/TP.0b013e3181b7ccc6. PMID 19935467
- [Background] Lin D, Hollander Z, Ng RT, Imai C, Ignaszewski A, Balshaw R, Freue GC, Wilson-McManus JE, Qasimi P, Meredith A, Mui A, Triche T, McMaster R, Keown PA, McManus BM; Biomarkers in Transplantation Team; NCE CECR Centre of Excellence for the Prevention of Organ Failure. Whole blood genomic biomarkers of acute cardiac allograft rejection. J Heart Lung Transplant. 2009 Sep;28(9):927-35. doi: 10.1016/j.healun.2009.04.025. PMID 19716046
- [Background] Kuzyk MA, Smith D, Yang J, Cross TJ, Jackson AM, Hardie DB, Anderson NL, Borchers CH. Multiple reaction monitoring-based, multiplexed, absolute quantitation of 45 proteins in human plasma. Mol Cell Proteomics. 2009 Aug;8(8):1860-77. doi: 10.1074/mcp.M800540-MCP200. Epub 2009 May 1. PMID 19411661
- [Derived] Lee H, Kovacs C, Mattman A, Hollander Z, Chen V, Ng R, Leung JM, Sin DD. The impact of IgG subclass deficiency on the risk of mortality in hospitalized patients with COPD. Respir Res. 2022 May 31;23(1):141. doi: 10.1186/s12931-022-02052-3. PMID 35641962
- [Derived] Takiguchi H, Chen V, Obeidat M, Hollander Z, FitzGerald JM, McManus BM, Ng RT, Sin DD. Effect of short-term oral prednisone therapy on blood gene expression: a randomised controlled clinical trial. Respir Res. 2019 Aug 5;20(1):176. doi: 10.1186/s12931-019-1147-2. PMID 31382977